CLINICAL TRIAL: NCT04917744
Title: Longitudinal Metabolite Levels in Patients Receiving Maintenance PARP Inhibitors
Brief Title: Metabolite Levels in Ovarian Cancer Patients Receiving Maintenance PARP Inhibitors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-013191; NCI-2021-02151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-013191 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (blood collection, chart review): Patients undergo collection of blood samples prior to drug initiation, weekly thereafter for the first month of therapy, monthly for the first month, and at disease progression or after cessation of treatment to monitor for toxicity. Blood samples are analyzed. Patients' medical charts are also reviewed to determine outcomes after PARP inhibition.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Laboratory Biomarker Analysis — Ancillary studies
Other: Medical Chart Review — Review of medical charts
  Other Names: Chart Review

SUMMARY:
This study evaluates blood samples and compares levels of metabolites (levels of vitamins, carbohydrates, proteins, etc., that are in the blood), before and after the plasma exchange in patients scheduled to receive immunotherapy for their ovarian cancer. The information gained from this study may help researchers better understand the side effects from each treatment and possibly lessen those side effects for future treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the extent to which PARP inhibitor (PARPi) treatment reduces systemic levels of mesenchymal stem cell (MSC)-derived cancer support factors in patients with cancer.

OUTLINE:

Patients undergo collection of blood samples prior to drug initiation, weekly thereafter for the first month of therapy, monthly for the first month, and at disease progression or after cessation of treatment to monitor for toxicity. Blood samples are analyzed. Patients' medical charts are also reviewed to determine outcomes after PARP inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with ovarian cancer starting PARP inhibitor treatment

Exclusion Criteria:

* Patients unwilling to return for blood draws, patients unwilling to continue PARP inhibitor treatment for at least one month

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with melanoma scheduled to receive immunotherapy for their ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Change of mesenchymal stem cell (MSC)-derived cancer support factors | At four weeks post PARP inhibitor treatment
  Levels of MSC-derived cancer support factors will be compared to baseline (i.e. pre-PARPi therapy) at each collection time point by Student's t test. In addition, outcomes by Cox proportional hazards will be compared between designated responders (i.e. patients whose MSC-derived cancer support factors decreased after PARP inhibition) and non-responders (i.e. patients whose MSC-derived cancer support factors did not decrease after PARP inhibition)

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years
  Stratified by extent of MSC-derived cancer support factor reduction. Will also compare levels at progression and/or after discontinuation of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J. Orme, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials